CLINICAL TRIAL: NCT00329914
Title: Effectiveness of Vaginally Administered Progesterone to Prevent Preterm Delivery in Twin Pregnancies - A Multicentre Randomized Trial
Brief Title: Does Progesterone Prevent Very Preterm Delivery in Twin Pregnancies?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Danish Medical Research Council (Other); The Danish Medical Society in Copenhagen (Unknown); AP Moeller Foundation (Other)
Responsible Party: Professor Ann Tabor, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: predict2006
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2009-02

CONDITIONS: Preterm Delivery
Keywords: Preterm delivery; Prevention; Twins; Progesterone
MeSH Terms: conditions — Premature Birth | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Progesterone (Active Comparator)
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — Vaginal pessaries, 200 mg/day
  Other Names: Utrogestan
  Arms: Progesterone
Drug: Placebo — Placebo pessaries containing peanut oil
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether a daily dose of 200 mg progesterone administered vaginally from 20-23 to 34 weeks' gestation will reduce the rate of preterm delivery amongst twin pregnancies.

DETAILED DESCRIPTION:
Multiple gestations account for 2% of all pregnancies, but cause more than 10% of the cases of preterm delivery. Due to increasing maternal age and use of assisted reproduction the number of multiple gestations is larger than ever. If markers of preterm delivery can be identified and means of preventing preterm delivery are found, it will be possible to reduce the number of children admitted to hospital because of prematurity.

Recently, two larger randomised studies investigated the effect of progesterone in singleton pregnancies of women who had previously delivered preterm. They both found a significant reduction in the preterm delivery rate in the progesterone group compared to a placebo group.

The study will be performed as a randomized, double-blind placebo controlled study of twin pregnancies in Denmark and Austria. The women will be randomised in a 1:1 ratio to two groups (progesterone versus placebo). Randomisation will be stratified per centre and according to chorionicity, as the risk of preterm delivery is doubled in monochorionic twins compared to dichorionic twins.

ELIGIBILITY:
Inclusion Criteria:

* Twin pregnancy
* Informed consent
* 18-23 weeks' gestation
* Participants must be fluent in the language spoken in the respective centres

Exclusion Criteria:

* Age < 18 years
* Known allergy to progesterone or peanuts
* Active thromboembolic disorders or a history of hormone-associated thromboembolic disorders
* Rupture of membranes at the time of inclusion
* Monoamniotic twins
* Pregnancies treated for or with signs of twin-to-twin transfusion syndrome at inclusion
* Multiple pregnancies reduced to twin pregnancies
* Known significant structural or chromosomal fetal abnormality
* Chorionicity not assessed before 15 weeks
* Known or suspected malignancy in genitals or breasts
* Known liver disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2006-06; Primary Completion 2009-02 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The incidence of delivery < 34 weeks, in the study group versus the control group | Participants will be followed until 3 weeks after delivery

SECONDARY OUTCOMES:
Physical and neurological development of the children at 6 and 18 months | 2 years after delivery
The relationship between cervical length and prophylactic progesterone treatment | Participants will be followed until 3 weeks after delivery
Determination of proteomics and RNA in preterm delivery and term delivery and an evaluation of the effect of progesterone on proteomics and RNA | Participants will be followed until 3 weeks after delivery
Assessment of the potential anti-inflammatory effect of progesterone by cytokine-measurements | Participants will be followed until 3 weeks after delivery
Assessment of the effect of progesterone on CRH-levels in twin pregnancies | Participants will be followed until 3 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Line Rode, MD, Principal Investigator — Ultrasound Clinic 4002, Rigshospitalet; Ann Tabor, professor, Study Director — Ultrasound Clinic 4002, Rigshospitalet
Locations (17):
- Austria (4):
  - Graz University Hospital, Graz
  - Innsbruck University Hospital, Innsbruck
  - Klagenfurt Hospital, Klagenfurt
  - Vienna University Hospital, Vienna
- Denmark (13):
  - Aalborg Hospital, Aalborg
  - Skejby Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Glostrup Hospital, Glostrup Municipality
  - Gentofte Hospital, Hellerup
  - Herlev Hospital, Herlev
  - Hilleroed Hospital, Hilleroed
  - Holbaek Hospital, Holbæk
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense
  - Roskilde Hospital, Roskilde
  - Soenderborg Hospital, Sønderborg
  - Viborg Hospital, Viborg

REFERENCES:
- [Result] Rode L, Klein K, Nicolaides KH, Krampl-Bettelheim E, Tabor A; PREDICT Group. Prevention of preterm delivery in twin gestations (PREDICT): a multicenter, randomized, placebo-controlled trial on the effect of vaginal micronized progesterone. Ultrasound Obstet Gynecol. 2011 Sep;38(3):272-80. doi: 10.1002/uog.9093. PMID 21739497
- [Result] Klein K, Rode L, Nicolaides KH, Krampl-Bettelheim E, Tabor A; PREDICT Group. Vaginal micronized progesterone and risk of preterm delivery in high-risk twin pregnancies: secondary analysis of a placebo-controlled randomized trial and meta-analysis. Ultrasound Obstet Gynecol. 2011 Sep;38(3):281-7. doi: 10.1002/uog.9092. PMID 21739499
- [Derived] Rode L, Klein K, Larsen H, Holmskov A, Andreasen KR, Uldbjerg N, Ramb J, Bodker B, Skibsted L, Sperling L, Hinterberger S, Krebs L, Zingenberg H, Weiss EC, Strobl I, Laursen L, Christensen JT, Skogstrand K, Hougaard DM, Krampl-Bettelheim E, Rosthoj S, Vogel I, Tabor A. Cytokines and the risk of preterm delivery in twin pregnancies. Obstet Gynecol. 2012 Jul;120(1):60-8. doi: 10.1097/AOG.0b013e31825bc3cd. PMID 22914392
- See also: Related Info — http://clinicaltrials.gov/ct2/show/NCT00329914